CLINICAL TRIAL: NCT05411081
Title: A Phase II Randomized Trial of Cabozantinib (NSC #761968) With or Without Atezolizumab (NSC #783608) in Patients With Advanced Papillary Renal Cell Carcinoma (PAPMET2)
Brief Title: Testing Cabozantinib With or Without Atezolizumab in Patients With Advanced Papillary Kidney Cancer, PAPMET2 Trial
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Other - CTEP request/poor accrual/pharma declined support
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-04668; NCI-2022-04668 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2200 (Other: SWOG); S2200 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2022-06-07; First posted 2022-06-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Papillary Renal Cell Carcinoma; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — atezolizumab; Specimen Handling; cabozantinib; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (cabozantinib S-malate) (Active Comparator): Patients receive cabozantinib S-malate PO QD on days 1-21 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan or MRI and blood and urine sample collection throughout the trial. Patients may also undergo bone scan throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Drug: Cabozantinib S-malate; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging
- Arm II (cabozantinib S-malate, atezolizumab) (Experimental): Patients receive cabozantinib S-malate PO QD on days 1-21 and atezolizumab IV over 30-60 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan or MRI and blood and urine sample collection throughout the trial. Patients may also undergo bone scan throughout the trial.
  Interventions: Biological: Atezolizumab; Procedure: Biospecimen Collection; Procedure: Bone Scan; Drug: Cabozantinib S-malate; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
  Arms: Arm II (cabozantinib S-malate, atezolizumab)
Procedure: Biospecimen Collection — Undergo collection of blood and urine samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scans
  Other Names: Bone Scintigraphy
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL 184; XL-184; XL184
Procedure: Computed Tomography — Undergo CT scans
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI

SUMMARY:
This phase II trial compares the effect of atezolizumab in combination with usual treatment with cabozantinib to cabozantinib alone in patients with papillary renal cell carcinoma that has spread from where it first started (primary site) to other places in the body (metastatic). Papillary renal cell carcinoma (PRCC) is a type of kidney cancer that forms in the lining of the tiny tubes in the kidney that return filtered substances that the body needs back to the blood and remove extra fluid and waste as urine. Most papillary tumors look like long, thin finger-like growths under a microscope. It is also called papillary kidney cancer or PRCC. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the tumor and may interfere with the ability of tumor cells to grow and spread. Cabozantinib is in a class of medications called kinase inhibitors. It works by blocking the action of an abnormal protein that signals tumor cells to multiply and may also prevent the growth of new blood vessels that tumors need to grow. By these actions it may help slow or stop the spread of tumor cells. Combination therapy with atezolizumab and cabozantinib may shrink the tumor and allow a longer survival time in patients with metastatic renal cell carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare progression-free survival in participants with metastatic papillary renal cell carcinoma (mPRCC) randomized to cabozantinib (cabozantinib S-malate) with atezolizumab versus cabozantinib alone.

SECONDARY OBJECTIVES:

I. To compare overall survival in participants with mPRCC randomized to cabozantinib with atezolizumab versus cabozantinib alone.

II. To compare Response Evaluation Criteria in Solid Tumors (RECIST) objective response rate (confirmed and unconfirmed, complete and partial response) in participants with mPRCC randomized to cabozantinib with atezolizumab versus cabozantinib alone.

III. To evaluate the quantitative and qualitive adverse events observed in each treatment arm.

BANKING OBJECTIVE:

I. To bank biospecimens for future correlative studies.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive cabozantinib S-malate orally (PO) once daily (QD) on days 1-21 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) and blood and urine sample collection throughout the trial. Patients may also undergo bone scan throughout the trial.

ARM II: Patients receive cabozantinib S-malate PO QD on days 1-21 and atezolizumab intravenously (IV) over 30-60 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan or MRI and blood and urine sample collection throughout the trial. Patients may also undergo bone scan throughout the trial.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a histologically confirmed diagnosis of metastatic papillary renal cell carcinoma (PRCC), either type 1 or type 2. (NOTE: A designation of type 1 or type 2 should be made by the local pathologist if possible but is not required). Mixed histologies which contain type 1 or type 2 along with any other RCC histology/histologies will be allowed provided that they contain a papillary component
* Participants must have measurable disease per RECIST 1.1 criteria. All measurable lesions must be assessed by CT or MRI within 28 days prior to registration. All non-measurable lesions must be assessed by CT or MRI, or nuclear medicine bone scan within 42 days prior to registration. The CT from a combined positron emission tomography (PET)/CT may be used to document only non-measurable disease unless it is of diagnostic quality. If there is clinical suspicion for bone metastases at the time of enrollment (at the discretion of the investigator), bone scan must be performed at baseline (within 42 days prior to registration)
* Participants with new or progressive brain metastases (active brain metastases) must not require immediate central nervous system (CNS) specific treatment at the time of study registration or anticipated during the first cycle of therapy. Patients with leptomeningeal disease are excluded from enrolling
* Participants with measurable disease, per RECIST version (v)1.1, must be present outside the CNS
* Participants must have no history of intracranial hemorrhage or spinal cord hemorrhage
* Participants must not have undergone stereotactic radiotherapy within 7 days prior to initiation of study treatment, whole-brain radiotherapy within 14 days prior to initiation of study treatment, or neurosurgical resection within 28 days prior to initiation of study treatment
* Participants must not have ongoing requirements for corticosteroids as therapy for CNS disease
* Participants, if needed, must receive a stable dose of anti-convulsant therapy
* Participants must not have cavitating pulmonary lesions
* Participants must not have uncontrolled pleural effusions, pericardial effusions, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Participants with indwelling catheters (e.g., PleurX [registered trademark]) are allowed
* Participants must not have tumor invading the gastrointestinal (GI) tract or evidence of endotracheal or endobronchial tumor within 28 days prior to registration
* Participants must not have evidence of tumor invading or encasing any major blood vessels
* Participants must not have had major surgery within 28 days prior to registration, and participants must have recovered from any adverse effects of surgery
* Participants must not have had prior treatment with cabozantinib for any reason
* Participants must not have had prior treatment or adjuvant therapy with PD-1/PD-L1 checkpoint inhibitors for any reason within the past 6 months
* Participants must not have received more than one prior systemic therapy for advanced or metastatic renal cell carcinoma with the exception of another VEGF inhibitor Food and Drug Administration (FDA)-approved for advanced RCC (i.e., pazopanib, bevacizumab, sorafenib or axitinib). If a participant develops metastatic disease within six months of discontinuation of adjuvant therapy, this will constitute one prior systemic therapy for advanced or metastatic RCC. If a patient develops metastatic disease and more than six months has elapsed since discontinuation of adjuvant therapy, this will not constitute prior systemic therapy for advanced or metastatic RCC
* Participants must not take within 14 days prior to registration, nor plan to take while on protocol treatment, any strong CYP3A4 inhibitors (e.g. boceprevir, cobicistat, danoprevir, elvitegravir/RIT, fluvoxamine, indinavir, itraconazole, ketoconazole, lopinavir/RIT, nefazodone, nelfinavir, posaconazole, ritonavir, telaprevir, telithromycin, tipranavir/RIT, or voriconazole,); Please refer to https://drug-interactions.medicine.iu.edu/MainTable.aspx for the updated CYP3A4 inhibitors or inducers
* Participants must not take within 14 days prior to registration, nor plan to take while on protocol treatment, any strong CYP3A4 inducers (e.g. avasimibe, phenytoin, rifampin, rifabutin); Please refer to https://drug-interactions.medicine.iu.edu/MainTable.aspx for the updated CYP3A4 inhibitors or inducers
* Participants must complete all prior radiation therapy at least 14 days prior to registration. Participants must have recovered to =< grade 1 from all associated toxicities at the time of registration unless the toxicity is determined to be not clinically significant by the registering investigator
* Participants must not be receiving or planning to receive any other investigational agents at time of registration
* Participants must not have been diagnosed with a clinically significant autoimmune disease, exceptions such as diabetes, eczema, and vitiligo are allowed. Other non-clinically significant autoimmune diseases are allowed if approved by the registering investigator
* Participants must not be on steroid doses > 10 mg prednisone equivalent. Replacement steroid doses for adrenal insufficiency will be allowed. Also, short duration steroid therapy to prevent allergic reactions are acceptable (e.g. prior to CT imaging)
* Participants must be >= 18 years of age
* Participants must have a complete physical examination and medical history within 28 days prior to registration
* Participants must have a Zubrod performance status of 0-2
* White blood count (WBC) >= 2 x 10^3/uL (within 28 days prior to registration)
* Absolute neutrophil count (ANC) >= 1.5 x 10^3/uL (within 28 days prior to registration)
* Platelet count >= 100 x 10^3/uL (within 28 days prior to registration)
* Lymphocyte count >= 0.5 x 10^3/uL (within 28 days prior to registration)
* Hemoglobin (>= 9 g/dL) (within 28 days prior to registration). Participants may be transfused to meet this criterion
* Total serum bilirubin =< 1.5 x the institutional upper limit of normal (ULN) unless history of Gilbert's disease (within 28 days prior to registration). Participants with history of Gilbert's disease must have total bilirubin =< 5 x institutional ULN
* Aspartate aminotransferase (AST) must be =< 3 x the institutional ULN unless the liver is involved with the tumor, in which case serum transaminase (SGOT) must be =< 5 x the institutional ULN (within 28 days prior to registration)
* Alanine aminotransferase (ALT), must be =< 3 x the institutional ULN unless the liver is involved with the tumor, in which case serum transaminase (SGPT) must be =< 5 x the institutional ULN (within 28 days prior to registration)
* Participants must have serum creatinine =< 2 x the institutional ULN OR creatinine clearance (either measured or calculated) > 30 mL/min and obtained within 28 days prior to registration
* Participants must not have any clinical evidence of congestive heart failure (CHF) (specifically, New York Heart Association [NYHA] class III [moderate] or class IV [severe]) at the time of registration
* Participants must not have known history of congenital long QT syndrome and must not have experienced unstable angina pectoris, clinically significant cardiac arrhythmias, or stroke (transient ischemic attack [TIA] or other ischemic event) within 90 days prior to registration
* Participants must not have experienced myocardial infarction or thromboembolic event requiring anticoagulation within 90 days of registration, unless clinically stable with ongoing medical management
* Participants must have urine protein < 3+ within 28 days prior to registration. If urine protein is 3+ or greater, then urine protein by 24-hour collection must show less than 3 grams of protein
* Participants must have documented blood pressure of systolic blood pressure (SBP) < 150 mm Hg or diastolic blood pressure (DBP) < 100 mm Hg within 14 days prior to registration
* Participants with known human immunodeficiency virus (HIV) must be on effective anti-retroviral therapy at registration and have undetectable viral load within 6 months of registration
* Participants with evidence of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load while on suppressive therapy within 6 months prior to registration, if indicated
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants currently being treated for HCV infection must have undetectable HCV viral load within 6 months prior to registration
* Participants must be able to take oral medications (i.e., swallow pills whole). Participants must not have gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures that could in the opinion of the treating investigator affect absorption, or active peptic ulcer disease. Participants with intractable nausea or vomiting are not eligible
* Participants must not have had any clinically-significant GI bleeding within 3 months prior to registration and participants must not have a GI disorder which (at the discretion of the investigator) bears a high risk of perforation or fistula (e.g. Crohn's disease)
* Participants must not have had hemoptysis of >= (2.5 mL) of red blood, and do not demonstrate any other signs indicative of pulmonary hemorrhage within 3 months prior registration
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Participants must not be pregnant or nursing, due to VEGF therapy being toxic to embryogenesis. Individuals who are of reproductive potential must have agreed to use an effective contraceptive method with details provided as a part of the consent process. A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen
* Participants must not be on warfarin, at therapeutic doses. Low dose aspirin for cardio-protection (per local applicable guidelines) and low molecular weight heparin (LMWH) are allowed
* Participants must be offered the opportunity to participate in specimen banking. With participant consent, specimens must be collected and submitted via the Southwest Oncology Group (SWOG) Specimen Tracking System
* Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines

  * NOTE: For participants with impaired decision-making capabilities, legally authorized representatives may sign and give informed consent on behalf of study participants in accordance with applicable federal, local, and Central Institutional Review Board (CIRB) regulations
* As a part of the OPEN registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause, assessed up to 5 years
  A proportional hazards model will be used to evaluate the experimental arm compared to the control arm, adjusted for the stratification factors as covariates in the model. A one-sided p-value =< 0.05 will indicate statistical significance. Participants last known to be alive and progression free are censored at date of last contact.

SECONDARY OUTCOMES:
Overall survival | From date of registration to date of death due to any cause, assessed up to 5 years
  Will be estimated by the Kaplan-Meier method, and a stratified log-rank test will be used to compare the treatment arms. Participants last known to be alive are censored at date of last contact.
Objective response rate | Up to 5 years
  Will be estimated to within +/- 11% (95% confidence interval).
Incidence of adverse events | Day 1 of each cycle
  Will be estimated to within +/- 11% (95% confidence interval). Will utilize the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 for toxicity and serious adverse event reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin L Maughan, Principal Investigator — SWOG Cancer Research Network
Locations (200):
- United States (200):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Mary Bird Perkins Cancer Center - Metairie, Metairie, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Touro Infirmary, New Orleans, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Duke Cancer Center Cary, Cary, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Farmington Health Center, Farmington, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm